CLINICAL TRIAL: NCT00672854
Title: Study Comparing a Soybean Oil-Based vs Olive Oil-Based Lipid Emulsion: Effects on Endothelial Function, Inflammatory Markers, Oxidative Stress, Immune Function,Insulin Sensitivity and Carb Metabolism Intensive Care Unit Patients
Brief Title: Study Comparing a Soybean Oil-Based With an Olive Oil-Based Lipid Emulsion in ICU Patients Requiring TPN
Acronym: TPN2
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Guillermo Umpierrez, MD, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00007587; TPN (Other Grant/Funding Number: Baxter Healthcare Corporation)
Record Dates: First submitted 2008-04-18; First posted 2008-05-06 (Estimated); Results first posted 2014-08-01 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-09

CONDITIONS: Parenteral Nutrition
Keywords: parenteral nutrition; lipid emulsion; nosocomial infection; mortality; endothelial function; inflammatory markers; oxidative stress; immune function; autonomic nervous system; insulin sensitivity; carbohydrate metabolism
MeSH Terms: conditions — Hyperphagia; Cross Infection; Insulin Resistance | interventions — ClinOleic; Fat Emulsions, Intravenous; soybean oil, phospholipid emulsion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intralipid 20% Intravenous Emulsion (Active Comparator): Subjects who require Total Parenteral Nutrition TPN receiving Intralipid 20% (soybean-based)
  Interventions: Drug: Intralipid, 20% Intravenous Emulsion
- ClinOleic 20% Intravenous Emulsion (Experimental): Subjects who require Total Parenteral Nutrition TPN receiving ClinOleic 20% (olive oil based)
  Interventions: Drug: ClinOleic 20% Intravenous Emulsion

INTERVENTIONS:
Drug: ClinOleic 20% Intravenous Emulsion — ClinOleic 20% is a lipid emulsion containing a mixture of refined olive oil (approximately 80%) and refined soybean oil (approximately 20%) corresponding to an essential fatty acid intake of approximately 20% of the total fatty acids intake.
  Other Names: Lipid Emulsion
  Arms: ClinOleic 20% Intravenous Emulsion
Drug: Intralipid, 20% Intravenous Emulsion — It is made up of 20% Soybean oil, 1.2% egg yolk phospholipids, 2.25% glycerin, and water for injection
  Other Names: 20% i.v. fat emulsion
  Arms: Intralipid 20% Intravenous Emulsion

SUMMARY:
Many hospitalized patients who are malnourished or not eating receive intravenous feeding or total parenteral nutrition (TPN). Despite improving nutrition, TPN may increase the risk of infections and hospital complications. We do not know why TPN increases hospital complications, but it may be caused by the high sugar or fat content in TPN solutions.

DETAILED DESCRIPTION:
This study compares the effect of a soybean oil-based versus an olive oil-based lipid emulsion in healthy volunteers and in critically ill patients. In healthy volunteers, your blood sugar levels, blood vessel function, and your ability to fight infections will be examined. In ICU patients, we examines whether use of the olive oil-based lipid emulsion may decrease the risk of infection and hospital complications.

ELIGIBILITY:
Inclusion criteria:

* Age: 18 - 80 years when initiating PN
* In medical/surgical ICU
* Has central venous access to administer PN
* Anticipated to receive PN ≥ 5 days

Exclusion criteria:

* Enrolled in an investigative study within the last 30 days prior to study entry
* Female patients: pregnant or breast feeding
* Has clinical sepsis (defined as mean arterial pressure (MAP) < 60 mmHg on ≥ 2 occasions and unstable BP despite pressor support) within 24 hours prior to study entry
* Has known cirrhosis or total bilirubin ≥ 10.0 mg/dL
* Has chronic renal failure (defined as requirement for hemodialysis or peritoneal dialysis therapy), or creatinine ≥ 3.5 mg/dL without continuous renal replacement therapy (CRRT), or requires acute post-operative dialysis
* Has an active malignancy (defined as requiring chemotherapy, radiation, and/or surgical intervention within 90 days prior to study entry) (excluding non-melanoma skin cancer)
* Has known AIDS
* Has a terminal illness (life expectancy < 7 days)
* Has undergone organ transplantation
* Has received PN with lipid within 48 hours prior to study entry
* Has mental disability to understand the scope and possible consequences of the study and the legally authorized representative is unavailable
* Has a baseline serum triglyceride > 400 mg/dL

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Umpierrez, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Grady Memorial Hospital, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia

REFERENCES:
- [Result] Umpierrez GE, Spiegelman R, Zhao V, Smiley DD, Pinzon I, Griffith DP, Peng L, Morris T, Luo M, Garcia H, Thomas C, Newton CA, Ziegler TR. A double-blind, randomized clinical trial comparing soybean oil-based versus olive oil-based lipid emulsions in adult medical-surgical intensive care unit patients requiring parenteral nutrition. Crit Care Med. 2012 Jun;40(6):1792-8. doi: 10.1097/CCM.0b013e3182474bf9. PMID 22488002

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at Grady Memorial Hospital, a major urban teaching hospital affiliated with Emory University and at Emory University Hospital, a tertiary referral academic institution in Atlanta, Georgia.
Pre-assignment Details: A total of 100 patients were randomized to either soybean oil-based (intralipid 20%) parenteral nutrition or olive oil-based (ClinOleic 20%) parenteral nutrition for up to 28 days. A total of 49 patients received soybean oil-based parenteral nutrition and a total of 51 patients received olive oil-based lipid emulsion in parenteral nutrition
Groups:
- Total Parenteral Nutrition (TPN) Given Intralipid 20%: TPN subjects receive Intralipid (soybean-based)
  Intralipid: TPN with Intralipid (20%)
- Total Parenteral Nutrition (TPN) Given ClinOleic 20%: TPN subjects receive ClinOleic 20% (olive oil based)
  ClinOleic: TPN with ClinOleic (20%)
Period: Overall Study
Arm/Group | Total Parenteral Nutrition (TPN) Given Intralipid 20% | Total Parenteral Nutrition (TPN) Given ClinOleic 20%
Started | 49 | 51
Completed | 49 | 51
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Total Parenteral Nutrition (TPN) Given Intralipid 20% | Total Parenteral Nutrition (TPN) Given ClinOleic 20% | Total
Number analyzed (Participants) | 49 | 51 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (15) | 46.4 (19) | 48.9 (17)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 35 | 71
  >=65 years | 13 | 16 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 23 | 45
  Male | 27 | 28 | 55

OUTCOME MEASURES:

1. Primary Outcome: Number of New Nosocomial Infections After 48 Hrs of Parenteral Nutrition (PN) Between the 2 Groups During Their Hospital Stay
Description: New nosocomial infections, defined as culture-proven infection including wound, drain, bloodstream, respiratory tract, and urinary tract infections during PN. The presence of nosocomial infections was diagnosed based on standardized Centers for Disease Control (CDC) guidelines for laboratory-confirmed bloodstream infection and did not distinguish catheter-related infections per se. The following daily information was evaluated by the study team for nosocomial infection surveillance: temperature (fever)curve, white blood cell counts, review of daily progress notes in the medical record, daily clinical microbiology laboratory culture data, orders for antimicrobial agents (agent, daily dose, and start/stop times will be recorded), review of all relevant dictated radiographic reports (e.g., chest radiographs, abdominal computer tomography), communication, as needed, with primary physicians and site infectious disease consultants, and use of the CDC guidelines.
Time Frame: 2 days after Parenteral Nutrition (up to 28 days post randomization)
Measure: Number; unit: number of nosocomial infections
Groups:
- Total Parenteral Nutrition (TPN) Given Intralipid 20%: Total Parenteral Nutrition (TPN) subjects receive Intralipid 20% (soybean-based)
  Intralipid: TPN with Intralipid (20%)
- Total Parenteral Nutrition (TPN) Given ClinOleic 20%: Total Parenteral Nutrition (TPN) subjects receive ClinOleic 20% (olive oil based)
  ClinOleic: TPN with ClinOleic (20%)
Arm/Group | Total Parenteral Nutrition (TPN) Given Intralipid 20% | Total Parenteral Nutrition (TPN) Given ClinOleic 20%
Number analyzed (Participants) | 49 | 51
number of nosocomial infections | 21 | 29

2. Secondary Outcome: Number of Days Patients Stayed in ICU During Parenteral Nutrition Between Treatment Groups
Description: The mean number of days patients stayed in the intensive care unit between the Intralipid 20% and ClinOleic 20% while they are on parenteral nutrition is calculated and compared
Time Frame: During Parenteral Nutrition (up to 28 days post randomization)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Total Parenteral Nutrition (TPN) Given Intralipid 20% | Total Parenteral Nutrition (TPN) Given ClinOleic 20%
Number analyzed (Participants) | 49 | 51
days | 15.2 (14) | 17 (18)

3. Secondary Outcome: Mean Plasma Concentration of C-reactive Protein in mg/L at Baseline, Day 3 and Day 7 Among the Treatment Groups Will be Measured
Description: Peripheral blood samples will be analyzed for circulating levels of inflammatory markers markers like plasma C-reactive protein (CRP) at baseline, day 3, and day 7 of soybean oil- and olive oil-based parenteral nutrition infusion and compared. A reading of less than 1 mg/L indicates low risk; a reading between 1 and 2.9 mg/L indicates intermediate risk; a reading greater than 3 mg/L indicates high risk and a reading above 10 mg/L indicates a need for further testing. Since the patients are sick and hospitalized, it is expected that their levels are elevated compared to normal subjects. The levels between the 2 groups are compared to see if there is any difference.Levels were measured in plasma using a solid phase, two-site sequential chemiluminescent immunometric assays on the Immulite analyzer.
Time Frame: Baseline, Day 3 and Day 7
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Total Parenteral Nutrition (TPN) Given Intralipid 20% | Total Parenteral Nutrition (TPN) Given ClinOleic 20%
Number analyzed (Participants) | 49 | 51
mg/L
  Baseline | 169.67 (125.05) | 152.45 (123.09)
  Day 3 | 109.48 (58.42) | 115.33 (66.80)
  Day 7 | 122.71 (80.68) | 146.63 (115)

4. Secondary Outcome: Mean Plasma Concentration of Tumor Necrosis Factor-alpha, in pg/mL is Measured Between the Two Treatment Groups
Description: Plasma concentration of circulating levels of inflammatory stress markers like tumor necrosis factor-alpha is measured at baseline, day 3, and day 7 among soybean oil- and olive oil-based parenteral nutrition infusion groups. The normal reference values are < or =2.8 pg/mL. Levels were measured in plasma using a solid phase, two-site sequential chemiluminescent immunometric assays on the Immulite analyzer.
Time Frame: Baseline, Day 3 and Day 7
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Total Parenteral Nutrition (TPN) Given Intralipid 20% | Total Parenteral Nutrition (TPN) Given ClinOleic 20%
Number analyzed (Participants) | 49 | 51
pg/mL
  Baseline | 0.12 (0.08) | 0.09 (0.03)
  Day 3 | 0.12 (0.05) | 0.09 (0.03)
  Day 7 | 0.10 (0.04) | 0.10 (0.07)

5. Secondary Outcome: Mean Change in Plasma Concentration of Cystine in Micromol Per Liter at Baseline, Day 3 and Day 7 Among the Treatment Groups
Description: Mean Plasma concentration of circulating levels of oxidative stress markers like levels of cystine at baseline, day 3, and day 7 are measured and compared between the soybean oil- and olive oil-based parenteral nutrition infusion groups. Levels were measured using iodoacetate to alkylate free thiols, derivatization with dansyl chloride to fluorescently tag amino groups, and high pressure liquid chromatography (HPLC) and fluorescence to separate, detect, and quantify the molecules.
Time Frame: Baseline, Day 3 and Day 7
Measure: Mean (Standard Deviation); unit: micromol per liter
Arm/Group | Total Parenteral Nutrition (TPN) Given Intralipid 20% | Total Parenteral Nutrition (TPN) Given ClinOleic 20%
Number analyzed (Participants) | 49 | 51
micromol per liter
  Baseline | 82.22 (43.74) | 75.8 (31.09)
  Day 3 | 88.65 (39.09) | 93.54 (36.04)
  Day 7 | 90.06 (42.28) | 87.7 (42.04)

6. Secondary Outcome: Mean Hospital Blood Glucose (mg/dL) in Diabetic Patients is Measured During Parenteral Nutrition Between the Two Treatment Groups
Description: Mean hospital blood glucose is measured as an indicator for insulin sensitivity. Capillary blood glucose was measured with a glucose meter at bedside during PN infusion. For this study normal blood glucose levels were indicated as 70-200 mg/dL, any blood glucose level < 70 mg/dL is regarded as hypoglycemia and above 200 mg/dL is regarded as hyperglycemia.
Time Frame: During Parenteral Nutrition (up to 28 days post randomization)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Total Parenteral Nutrition (TPN) Given Intralipid 20% | Total Parenteral Nutrition (TPN) Given ClinOleic 20%
Number analyzed (Participants) | 49 | 51
mg/dL | 128.4 (6) | 125 (9)

7. Secondary Outcome: Number of Deaths During Parenteral Nutrition Treatment Between Two Treatment Groups During Hospitalization
Description: Mortality is defined as death occurring during admission, either during the time PN is received or after PN treatment is completed. Death during hospitalization rather than during PN treatment was chosen because many patients who undergo treatment with PN die or develop hospital complications within a period of several days after treatment cessation. The number of deaths between the two groups are compared.
Time Frame: During Parenteral Nutrition (up to 28 days post randomization)
Measure: Number; unit: participants
Arm/Group | Total Parenteral Nutrition (TPN) Given Intralipid 20% | Total Parenteral Nutrition (TPN) Given ClinOleic 20%
Number analyzed (Participants) | 49 | 51
participants | 5 | 4

8. Secondary Outcome: Mean Change in Percentage of Granulocyte Phagocytosis After 7-day Administration of Parenteral Nutrition Between the Two Treatment Groups
Description: Change in immune function is assessed by percentage of Granulocyte phagocytosis after 7-day administration of parenteral nutrition between the two treatment groups. The phagocytic and oxidative burst activity of monocytes and granulocytes in heparinized whole blood was assessed according to manufacturer's instructions using specific reagent kits for this purpose at baseline and again at day 7. Briefly, granulocyte phagocytic activity was quantitated by incubation of whole blood with fluorescein isothiocyanate-labeled, opsonized Escherichia coli bacteria at 37°C with detection of fluorescence of internalized particles as a percentage of positive cells by flow cytometry.
Time Frame: Baseline and 7 days post randomization
Measure: Mean (Standard Deviation); unit: percentage of phagocytosis
Arm/Group | Total Parenteral Nutrition (TPN) Given Intralipid 20% | Total Parenteral Nutrition (TPN) Given ClinOleic 20%
Number analyzed (Participants) | 49 | 51
percentage of phagocytosis | 3.86 (18.8) | 6.36 (38.4)

ADVERSE EVENTS:
Time Frame: The adverse events were calculated up to 28 days post randomization and on parenteral nutrition between the two treatment groups
Description: Since the subjects enrolled are already hospitalized patients in the Intensive care unit, main adverse events of interest were serious adverse events and deaths are captured for the study
Groups:
- Total Parenteral Nutrition (TPN) Given Intralipid 20%: TPN subjects receive Intralipid 20% (soybean-based)
  Intralipid: TPN with Intralipid (20%)
Arm/Group | Total Parenteral Nutrition (TPN) Given Intralipid 20% | Total Parenteral Nutrition (TPN) Given ClinOleic 20%
All-Cause Mortality (participants affected / at risk) | 5/49 | 4/51
Serious Adverse Events (participants affected / at risk) | 33/49 | 44/51
Other Adverse Events (participants affected / at risk) | 2/49 | 3/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Total Parenteral Nutrition (TPN) Given Intralipid 20% (N=49) | Total Parenteral Nutrition (TPN) Given ClinOleic 20% (N=51)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Urinary tract infection, (Renal and urinary disorders) | 7 | 7
Bacteremia (Blood and lymphatic system disorders) | 11 | 11
Wound infection, (Skin and subcutaneous tissue disorders) | 4 | 11
Acute myocardial infarction, (Cardiac disorders) | 0 | 2
Congestive heart failure, (Cardiac disorders) | 1 | 2
Cardiac arrhythmia, (Cardiac disorders) | 5 | 6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Total Parenteral Nutrition (TPN) Given Intralipid 20% (N=49) | Total Parenteral Nutrition (TPN) Given ClinOleic 20% (N=51)
Vein irritation (Surgical and medical procedures) | 2 | 3

LIMITATIONS AND CAVEATS:
Limitations of the study included the relatively small number of patients, the preponderance of surgical ICU subjects, and that the study was not powered to demonstrate differences in mortality between treatment groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No